CLINICAL TRIAL: NCT04456608
Title: Program on Genetic and Dietary Predictors of Drug Response in Rural and AI/AN Populations, Project-3, SA-3, Anti-platelet Response
Brief Title: Genetic and Dietary Predictors of Anti-platelet Response
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding ended before the study could be completed,
Sponsor: University of Washington (Other)
Collaborators: Southcentral Foundation (Other); University of Montana (Other); Oregon Health and Science University (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Kenneth Thummel, Professor: Pharmaceutics, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SITE00000212; 5P01GM116691 (NIH)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Platelet Function
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: In this study we will recruit individuals who have previously been determined to have low or high RBC n-3 PUFA content and test platelet function at baseline and after 2-day aspirin treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Low and High n-3 PUFA (Experimental): Individuals with low or high n-3 PUFA RBC concentration will be given aspirin (81 mg of aspirin once a day, for 6 days)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Low and high n-3 PUFA participants will receive 81-mg aspirin once a day, for 6 days.

SUMMARY:
This study will investigate differences in platelet aggregation under basal and aspirin-treated conditions in American Indian and Alaska Native people who have extreme levels (low and high) of n-3 polyunsaturated fatty acids (n-3 PUFAs, EPA and DHA) in red blood cell membranes. The study will also determine whether or not platelet aggregation under the different conditions is modified by CYP4A11, CYP4F2, CYP4F11, PEAR1, and ACTN1 gene variation.

DETAILED DESCRIPTION:
Purpose: In this aim, the investigators will test the hypothesis that n-3 PUFAs modify aspirin anti-platelet response, by measuring and comparing three different indicators of aspirin response in individuals with extremely high and low RBC n-3 PUFA levels, under a basal state and after 1-week of once a day aspirin treatment. The three indicators are: 1) platelet TXB2 and 20-HETE concentrations; 2) platelet aggregation ex vivo (in response to external stimuli); and 3) aspirin covalent adduct of COX-1. The investigators will also test whether or not common variants in the CYP4A11, CYP4F2, CYP4F11, PEAR1 and ACTN1 genes are associated with basal and aspirin-induced changes in platelet aggregation and, in an exploratory analysis, modify the effects of n-3 PUFAs on aspirin response.

Procedures and Population: Investigators from the University of Montana, Southcentral Foundation and Oregon Health & Science University will recruit a total of 150 individuals (50 at each site) to participate in the study. At each performance site, the participants recruited will represent 25 individuals with high and 25 individuals with low RBC n-3 PUFA concentrations. After providing written consent, each study participant will be screened for medical history and clinical lab testing to ensure good health and good liver, kidney and blood test parameters. If found to be eligible, each participant will provide 12-hour fasted (overnight) blood samples for isolation of plasma, platelets, lymphocytes, and red blood cells. A separate blood sample will be collected into a citrate treated tube for platelet aggregation testing using the PFA-100 platform. Isolated blood fractions will be stored at -80°C.

After baseline sampling, each participant will be given six doses of aspirin (80 mg/day for 2 days) and instructed to take one dose daily at approximately 9 am. On the day after the last aspirin dose, the participant will provide blood samples for repeated platelet aggregation testing, platelet lipid analysis and measurement of aspirin covalent adduct to COX-1, and a spot urine sample to confirm aspirin consumption by testing for salicylate. For 24 hours prior to platelet aggregation testing, study participants will be asked to avoid foods that could lead to spurious test results (eg, chocolate, tea, coffee, cola, red wine, beer, tomato, grapes, grape juice, orange and cranberry juices, as well as traditional wild foods that include berries, plant roots, plant greens etc).

Analytical Methods: Whole blood, point of care, platelet aggregation testing will be performed using the automated PFA-100 instrument. Performance by research personnel will be compared head-head to clinical testing services at each site, as a quality control measure. In each test setting, the investigators will obtain results in duplicate for both collagen/epinephrine and collagen/ADP cartridges. The investigators will also measure platelet TXB2, 20-HETE and AA concentrations, by LC-MS/MS. In addition, the investigators will develop and employ a method to quantify theaspirin covalent adduct of COX-1 in isolated platelets from study participants.

Statistical Methods: For each study population, and subgroups with extreme RBC n-3 PUFA phenotypes, the investigators will use linear regression models with robust standard errors to identify significant differences in the mean absolute platelet aggregation test results under basal and aspirin-treated conditions (primary outcome), as well as the post-treatment-to-baseline change in platelet aggregation. Heterogeneity between pairs of extreme phenotypes subgroups will be accounted for by including sex, age, BMI and platelet count as covariates in the regression model. Sample size calculation for each performance site (n = 25 per n-3 PUFA subgroup) was based on having power of at least 0.8 for detecting a difference in mean platelet aggregation between the two extreme (0-10 and 90-100 percentiles) n-3 PUFA subgroups under basal conditions, at a significance level of 0.05. As a secondary level of analysis, for each subgroup of the extreme RBC n-3 PUFA phenotypes, the investigators will also compare mean platelet TXB2 and 20-HETE concentrations under basal and aspirin-treated conditions, as well as the post-treatment-to-baseline change. Finally, a third level of analysis will involve testing each study population for a difference in the extent of aspirin adduct to COX-1 between groups with extreme RBC n-3 PUFA phenotypes. The investigators will test for associations between platelet aggregation test results and biochemical measures of platelet activation, each study population separately and in aggregate.

The investigators will use linear regression models to test for an association between common CYP4A11,CYP4F2, CYP4F11, PEAR1 and ACTN1 genotypes and the mean absolute platelet aggregation test results under basal and aspirin-treated conditions, as well as the post-treatment-to-baseline change in platelet aggregation. In an exploratory analysis, the investigators will apply Linear Mixed Effects (LME) models to the combined pre- and post-treatment dataset to test for associations with n-3 PUFAs group and drug effects, as well as to identify any modifications of those effects by CYP4A11, CYP4F2, CYP4F11, PEAR1 and ACTN1 variation by including and testing for significant interaction effects in the models. The investigators will include random effects in the LME to account for potential heterogeneity in each of the populations.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with no history of significant medical conditions including cardiac, pulmonary, hepatic, gastrointestinal, or renal disease, or HIV.
2. Participants will be males or females, 18 years or older.
3. Participants will be self-identified as: Yup'ik or Cup'ik (YK-Delta), AI/AN (SCF), or a member of the Confederated Salish and Kootenai Tribe (Flathead Reservation).
4. Participants must read and understand English or Yup'ik.
5. Participants must be able to provide informed consent.

Exclusion Criteria:

1. Participants with any significant chronic medical condition, including cardiac, pulmonary, hepatic, gastrointestinal, or renal disease, or HIV.
2. Participants less than 18 yrs of age.
3. Participants unable to read and understand English or Yup'ik.
4. Participants unable to provide informed consent.
5. Recent (within 2 weeks) use of aspirin, NSAIDs, antihistamines, or any prescription anticoagulant drug such as warfarin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
PFA-100 Platelet Aggregation Test | Single 9 am blood sample on day 3 of study
  Citrated blood samples will be treated with collagen/epinephrine and collagen/ADP and the time to reach an aggregation endpoint will be measured.

SECONDARY OUTCOMES:
Platelet TBX2 concentration | Single 9 am blood sample on day 3 of study
  Platelet TBX2 concentration
Platelet 20-HETE concentration | Single 9 am blood sample on day 3 of study
  Platelet 20-HETE concentration

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth E Thummel, Ph.D., Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - Southcentral Foundation, Anchorage, Alaska
  - University of Montana, Missoula, Montana
  - Oregon Health & Sciences University, Portland, Oregon